CLINICAL TRIAL: NCT06649721
Title: Innovating Shorter, All- Oral, Precised Treatment Regimen for Rifampicin Resistant Tuberculosis：BDLL Chinese Cohort
Acronym: INSPIRE-BDLL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Head of Infectious Disease Department, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSPIRE-BDLL
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Drug-resistant Tuberculosis; Pulmonary Tuberculosis; Rifampin-resistant Tuberculosis
Keywords: Drug-resistant tuberculosis; BDLL; Chinese Population; Short regimen
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis, Pulmonary | interventions — bedaquiline; OPC-67683; Fumigant 93; Linezolid; Levofloxacin; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BDLL (Experimental): 6-month all-oral regimen, consisting of Bedaquiline (BDQ, B), Delamanid (DLM, D), Linezolid (LZD, L), Levofloxacin (LFX) or Clofazimine (CFZ, C), as known as BDLLfxC or BDLL regimen
  Interventions: Drug: bedaquiline; Drug: delamanid; Drug: linezolid; Drug: Levofloxacin; Drug: Clofazimine

INTERVENTIONS:
Drug: bedaquiline — 400 milligrams (mg) daily for 2 weeks(w), then 200mg three times a week for 22 weeks (w)
  Other Names: BDQ; B
Drug: delamanid — * for participants weighing up to 33.9 kilograms (kg): 50mg two times a day for 24w
  * for participants weighing 34kg or above: 100mg two times a day for 8w, then 200mg daily for 16w
  Other Names: DLM; D
Drug: linezolid — * for participants weighing up to 33.9kg: 450mg daily;
  * for participants weighing 34kg or above: 600mg daily; for 24w if a negative culture is obtained from sputum collected at 16w, or else for 36w
  Other Names: LZD; L
Drug: Levofloxacin — Only for participants with confirmed fluoroquinolone-susceptible TB or unknown fluoroquinolone susceptibility:
  * for participants weighing up to 33.9kg: 500mg daily
  * for participants weighing 34kg to 49.9kg: 750 daily
  * for participants weighing 50kg or above: 1000mg daily for 24w if a negative culture is obtained from sputum collected at 16w, or else for 36w
  Other Names: LFX
Drug: Clofazimine — Only for participants with confirmed fluoroquinolone-resistant TB or unknown fluoroquinolone susceptibility:
  100mg daily, for 24w if a negative culture is obtained from sputum collected at 16w, or else for 36w
  Other Names: CFZ; C

SUMMARY:
This is an investigational, prospective, multicenter, single-arm, open label trial. The goal of this clinical trial is to evaluate the efficacy and safety of a 6-month all-oral regimen, consisting of Bedaquiline (BDQ, B), Delamanid (DLM, D), Linezolid (LZD, L), Levofloxacin (LFX) or Clofazimine (CFZ, C), or BDLLfxC regimen, to treat rifampin-resistant pulmonary tuberculosis (RR-TB) in Chinese teenagers and adults (aged 12 years or above). The main questions it aims to answer are:

* Is BDLLfxC regimen effective to treat RR-TB in Chinese participants?
* Is BDLLfxC regimen safe in Chinese RR-TB participants? Participants will take BDLLfxC regimen to treat their RR-TB. There will be no additional hospital visits, laboratory tests or radiological examinations other than routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing to sign informed consent of this trial, those without capacity for civil conduct need their legal guardian to sign
* Participants (and their legal guardian if applicable) are willing to cooperate to complete all trial procedures
* Male or female, 12 years or older, weight ≥ 30kg
* Confirmed pulmonary tuberculosis with resistance to rifampin by phenotypic or genotypic susceptibility testing within 3 months, and must be re-confirmed by sputum culture sampled at trial inclusion
* Women with childbearing potential should not be pregnant, confirmed by a volunteered negative pregnancy test, and are willing to use effective contraceptive method from giving consent to 3 months after study treatment
* Men with childbearing potential must be willing to use condom or other effective contraceptive methods to avoid their sex partners from being pregnant
* Women in breastfeeding period must be willing to discontinue breastfeeding from giving consent to 3 months after study treatment
* Participants are willing to take HIV test, and willing to take appropriate antiretroviral therapy if positive

Exclusion Criteria:

* Previously use of Bedaquiline or Delamanid for at least 28 days
* Concomitant hematogenous disseminated tuberculosis, or severe pulmonary tuberculosis in investigator's opinion (including tuberculosis of the digestive system, osteoarticular tuberculosis or tuberculous meningitis)
* Currently using any drug that has been prohibited in the protocol
* History of allergic action to any of the study drugs
* Currently participating in any other clinical trials
* Cardiovascular risk at screening: (1) QTcF more than 480 milliseconds (ms); (2) History of clinically significant arrythmia, and at investigator's opinion, participation in this study will increase the risk; (3) Decompensated heart failure; (4) Grade 3 high blood pressure and the goals of treatment have not been reached; (5) Abnormal thyroid function; (6) Abnormal serum Ca, Mg or K level; (7) Other conditions with cardiovascular risks in investigator's opinion.
* History of optic neuropathy or peripheral neuropathy, and the investigator considers that the condition may progress or deteriorate by participating in the study, or inappropriate to participate
* Hepatic disorders at screening: (1) Active viral hepatitis: HBsAg positive or HBV DNA >1000 CPs/mL, with elevated AST or ALT or HCV RNA positive; (2) Decompensated cirrhosis
* Renal disorders at screening: (1) Unstable or rapidly progressive renal disease; (2) Moderate / severe renal disfunction or end-stage renal disease (eGFR< 60 mL/min/1.73 m2); (3) Serum creatinine ≥133 μmol/L(1.5 mg/mL) in men, or ≥124 μmol/L (1.4 mg/mL) in women
* Other abnormal laboratory test: (1) Hemoglobin < 8.0g/dL; (2) Platelet <75,000/mm3; (3) Absolute neutrophil count <1000/mm3; (4) Aspartate transaminase (AST) or alanine aminotransferase (ALT) >3×upper limit of normal (ULN); (5) Total bilirubin (TBil) >2×ULN, or >1.5×ULN together with abnormal AST or ALT; (6) Albumin <30g/L
* The investigator considers that the participant is not able to complete the study process, or the participation is not safe.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with favorable outcomes in both treatment and follow-up period | Up to 72 weeks after start of treatment
  Favorable outcome in treatment period (up to 28 weeks after start of treatment): a participant's outcome will be defined as "favorable" if it meets any of the following below and has not been defined as "unfavorable" before,
  1. . Cured: complete at least 80% of total required dose per protocol, with negative culture results of last two sputum samples (collected 14 days apart) ;
  2. . Treatment completed: complete at least 80% of total required dose per protocol, with NO negative culture results of last two sputum samples (collected 14 days apart); Favorable outcome in follow-up period (from end of treatment to 72 weeks after start of treatment): a participant's outcome will be defined as "favorable" if it meets any of the following below and has not been defined as "unfavorable" before,
  (1). Cured: sputum culture negative at 72 weeks from start of treatment; (2). Culture negative when last seen: loss to follow-up before 72 weeks, with negative sputum culture when last seen.

SECONDARY OUTCOMES:
Proportion of participants with grade 3 or 4 adverse effect | Up to 72 weeks after start of treatment
  Adverse effect will be graded using Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Proportion of participants with favorable outcomes in treatment period, follow-up period and prolonged follow-up period, respectively | Up to 108 weeks after start of treatment
  The definitions of favorable outcome in treatment and follow-up period are as described in primary outcome. Favorable outcome in prolonged follow-up period (from end of treatment to 108 weeks after start of treatment): a participant's outcome will be defined as "favorable" if it meets any of the following below and has not been defined as "unfavorable" before, (1). Cured: sputum culture negative at 108 weeks from start of treatment; (2). Culture negative when last seen: loss to follow-up before 108 weeks, with negative sputum culture when last seen.
Time to culture conversion | Up to 72 weeks after start of treatment
  Time from start of treatment to the first time that obtained two consecutive negative sputum culture results, and the sputum samples must be collected 14 days apart. The date when first sputum sample is collected will be recorded as the date for culture conversion.

CONTACTS AND LOCATIONS:
Locations (34):
- China (34):
  - Anhui Chest Hospital, Hefei, Anhui
  - The 8th Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Fourth People's Hospital of Nanning, Nanning, Guangxi
  - Liupanshui Third People's Hospital, Liupanshui, Guizhou
  - Hebei Chest Hospital, Shijiazhuang, Hebei
  - The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - Infectious Disease Hospital of Heilongjiang Province, Harbin, Heilongjiang
  - Jiamusi Tuberculosis Hospital(Jiamusi Cancer Hospital), Jiamusi, Heilongjiang
  - Harbin Chest Hospital, Harbin, Helongjiang
  - Luoyang Center Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Chest Hospital, Zhengzhou, Henan
  - Henan Infectious Disease Hospital, Zhengzhou, Henan
  - Wuhan Pulmonary Hospital，Wuhan Tuberculosis Prevention and Control Institute, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Hulunbuir Infectious Disease Hospital, Hulunbuir, Inner Mongolia
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Jiangxi Chest Hospital, Nanchang, Jiangxi
  - Infectious Disease Hospital of Changchun, Changchun, Jilin
  - Jilin Tuberculosis Hospital, Jilin, Jilin
  - Shenyang Chest Hospital, Shenyang, Liaoning
  - Xi'an Chest Hospital, Xi'an, Shaanxi
  - Shandong Public Health Clinical Center, Shandong University, Jinan, Shandong
  - Linyi People Hospital, Linyi, Shandong
  - Qingdao Chest Hospital, Qingdao, Shandong
  - Weifang No.2 People's Hospital, Weifang, Shandong
  - Yantai Qishan Hospital, Yantai, Shandong
  - Shanxi Medical University Affiliated Chest Hospital, Taiyuan, Shanxi
  - Public Health Clinical Center of Chengdu, Chengdu, Sichuan
  - Tianjin Haihe Hospital, Tianjin, Tianjin Municipality
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - Beijing Chest Hospital, Beijing
  - Huashan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No